CLINICAL TRIAL: NCT01190813
Title: A Randomized Trial of Levodopa as Treatment for Residual Amblyopia (ATS 17)
Brief Title: Levodopa for the Treatment of Residual Amblyopia
Acronym: ATS17
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATS 17; 2U10EY011751 (NIH)
Record Dates: First submitted 2010-08-17; First posted 2010-08-30 (Estimated); Results first posted 2015-02-13 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Amblyopia
Keywords: amblyopia, levodopa
MeSH Terms: conditions — Amblyopia | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levodopa/Carbidopa (Active Comparator): Levodopa 0.76 mg/kg with Carbidopa 0.17 mg/kg tid
  Interventions: Drug: Levodopa/Carbidopa; Other: Patching
- Placebo (Placebo Comparator): Oral placebo tid
  Interventions: Drug: Placebo; Other: Patching

INTERVENTIONS:
Drug: Levodopa/Carbidopa — Oral levodopa 0.76 mg/kg tid with carbidopa 0.17 mg/kg tid
  Arms: Levodopa/Carbidopa
Drug: Placebo — Oral placebo tid
  Arms: Placebo
Other: Patching — Two hours of daily patching

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of oral levodopa and patching versus oral placebo and patching as treatment for residual amblyopia in children 7 to <13 years old with visual acuity of 20/50 to 20/400 in the amblyopic eye.

DETAILED DESCRIPTION:
Amblyopia is the most common cause of monocular visual impairment in both children and young and middle-aged adults. Both patching and atropine are accepted treatment modalities for the management of moderate amblyopia in children. Despite best efforts with conventional amblyopia treatment, many older children and teenagers with amblyopia fail to achieve normal visual acuity in the amblyopic eye. In a previous PEDIG study where children 7 to 12 years old were treated with atropine and patching, only 36% of the children with moderate amblyopia and only 23% of the children with severe amblyopia achieved 20/40 or better acuity.

Many clinicians have recognized that conventional therapies with patching and atropine have not been universally successful and have sought alternatives. PEDIG has discussed for several years the problem of residual amblyopia and how the remaining visual acuity deficit could be reduced. A number of research groups have evaluated the short term use of oral levodopa-carbidopa as an adjunct to patching therapy for older children.

ELIGIBILITY:
Inclusion Criteria:

1. Age 7 to 12
2. Amblyopia associated with strabismus, anisometropia, or both

   * Criteria for strabismus: One of the following criteria must be met: Heterotropia at distance and/or near fixation on examination (with or without spectacles); History of strabismus surgery; Documented history of strabismus which is no longer present (which in the judgment of the investigator could have caused amblyopia)
   * Criteria for anisometropia: One of the following criteria must be met: ≥0.50 D difference between eyes in spherical equivalent; ≥1.50 D difference between eyes in astigmatism in any meridian
3. Visual acuity, measured in each eye (amblyopic eye without cycloplegia) within 7 days prior to enrollment using the E-ETDRS protocol by a study certified visual acuity tester as follows:

   * Visual acuity in the amblyopic eye 18 to 67 letters inclusive (20/50 to 20/400)
   * Visual acuity in the fellow eye ≥78 letters (20/25 or better)
4. Current amblyopia treatment (other than spectacles)

   * 12 weeks of at least 2 hours of occlusion per day prescribed for the fellow eye during the immediate pre-enrollment period.
   * While on current treatment, visual acuity has not improved one line (5 letters) or more since a non-study visit at least 6 weeks ago. Both acuity measurements to define no improvement must have been done using the same testing method.
   * Treatment with atropine at any time during this pre-enrollment period is not allowed.
   * Any treatment prior to the current patching episode with stable acuity is acceptable.
5. Spectacle correction (if applicable) for measurement of enrollment visual acuity must meet the following criteria and be based on a cycloplegic refraction that is no more than 6 months old:

   1. Requirements for spectacle correction:

      * Spherical equivalent must be within 0.50 D of fully correcting the anisometropia.
      * Hypermetropia of 3.00D or more must be corrected.
      * Hypermetropia must not be under corrected by more than 1.50 D spherical equivalent, and reduction in plus sphere must be symmetric in the two eyes.
      * Cylinder power in both eyes must be within 0.50 D of fully correcting the astigmatism.
      * Cylinder axis in both eyes is within 6 degrees of the axis in the spectacles when cylinder power is ≥1.00 D.
      * Myopia of amblyopic eye greater than 0.50 D by spherical equivalent must be corrected, and the glasses must not under correct the myopia by more than 0.25 D or overcorrect it by more than 0.50 D.
   2. Spectacles meeting above criteria must be worn :until visual acuity in amblyopic eye is stable (defined as 2 consecutive visual acuity measurements by the same testing method at least 4 weeks apart with no improvement of one line (5 letters) or more.
6. Eye examination within 6 months prior to enrollment
7. Parent available for at least one year of follow-up, has access to phone), and willing to be contacted by clinical site and Jaeb Center staff
8. In the investigator's judgment, the subject is likely to comply with prescribed treatment (e.g., no history of poor compliance with patching treatment) and unlikely to continue to improve by using 2 hours of patching per day alone.

Exclusion Criteria:

1. Myopia more than -6.00 D (spherical equivalent) in either eye.
2. Current vision therapy or orthoptics
3. Ocular cause for reduced visual acuity

   * nystagmus per se does not exclude the subject if the above visual acuity criteria are met
4. Prior intraocular or refractive surgery
5. History of narrow-angle glaucoma
6. Bronchial asthma or severe pulmonary disease
7. Strabismus surgery planned within 26 weeks
8. Known allergy to levodopa or carbidopa
9. History of dystonic reactions
10. Current use of oral iron supplements including multivitamins containing iron during treatment with levodopa-carbidopa
11. Current use of antihypertensive, anti-depressant medications, phenothiazines, butyrophenones, risperidone and isoniazid, non-specific monoamine oxidase inhibitors, or medication for the treatment of attention deficit hyperactivity disorder
12. Known liver disease
13. History of melanoma
14. Known psychological problems
15. Known skin reactions to patch or bandage adhesives
16. Prior levodopa treatment
17. Treatment with topical ophthalmic atropine within the past 12 weeks
18. A physician-prescribed diet high in protein
19. Females who are pregnant, lactating, or intend to become pregnant within the next 34 weeks.

    * A negative urine pregnancy test will be required for all females who have experienced menarche.
    * Requirements regarding pregnancy testing prior to enrollment may be further defined by each individual Institutional Review Board.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 139 (Actual)
Dates: Start 2010-09; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael X Repka, MD, Study Chair — Jaeb Center for Health Research
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset is available on the PEDIG public website at http://pedig.jaeb.org/Studies.aspx?RecID=196

REFERENCES:
- [Result] Pediatric Eye Disease Investigator Group; Repka MX, Kraker RT, Dean TW, Beck RW, Siatkowski RM, Holmes JM, Beauchamp CL, Golden RP, Miller AM, Verderber LC, Wallace DK. A randomized trial of levodopa as treatment for residual amblyopia in older children. Ophthalmology. 2015 May;122(5):874-81. doi: 10.1016/j.ophtha.2015.01.002. Epub 2015 Feb 9. PMID 25676904
- See also: PubMed abstract — http://www.ncbi.nlm.nih.gov/pubmed/25676904
- See also: PubMed Central HHS Public Access - Full Text — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4414716/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2010 and October 2013, 139 participants from 27 sites were randomly assigned to levodopa (n=90) or placebo (n=49).
Period: Overall Study
Arm/Group | Levodopa/Carbidopa | Placebo
Started | 90 | 49
2-week Phone Call | 87 (2 missed, 1 dropped) | 48 (1 missed, 0 dropped)
4-week Visit | 88 (0 missed, 1 dropped) | 47 (1 missed, 1 dropped)
7-week Phone Call | 85 (3 missed, 0 dropped) | 46 (2 missed, 0 dropped)
10-week Visit | 88 (0 missed, 0 dropped) | 48 (0 dropped, 0 missed)
13-week Phone Call | 82 (6 missed, 0 dropped) | 48 (0 dropped, 0 missed)
16-week Visit | 87 (1 dropped) | 46 (2 dropped)
18-week Visit (Masked Primary) | 87 (0 dropped) | 45 (1 dropped)
23-week Phone Call | 82 (4 missed, 1 dropped) | 41 (4 missed, 0 dropped)
26-week Visit | 86 (0 missed, 0 dropped) | 45 (0 missed, 0 dropped)
Completed | 86 | 45
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Refused study treatment after randomized | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levodopa/Carbidopa | Placebo | Total
Number analyzed (Participants) | 90 | 49 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 90 | 49 | 139
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.4 (1.8) | 9.5 (1.7) | 9.5 (1.7)
Age, Customized [Number; unit: participants]
  7 to <9 years | 39 | 21 | 60
  9 to <11 years | 33 | 14 | 47
  11 to <13 years | 18 | 14 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 24 | 64
  Male | 50 | 25 | 75
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 1 | 3
  Black/African American | 1 | 1 | 2
  Hispanic or Latino | 5 | 2 | 7
  White | 77 | 44 | 121
  Unknown/Not Reported | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 90 | 49 | 139
Cause of Amblyopia [Number; unit: participants]
  Strabismus | 22 | 5 | 27
  Anisometropia | 20 | 16 | 36
  Combined Mechanism | 48 | 28 | 76
Patching Duration at Randomization [Number; unit: participants]
  2 hours per day | 81 | 43 | 124
  >= 3 hours per day | 9 | 6 | 15
Visual Acuity in the Amblyopic Eye at Randomization [Number; unit: participants]
  20/200 or worse (<=37 letters) | 7 | 9 | 16
  20/100 to <20/200 (38-52 letters) | 34 | 13 | 47
  20/80 (53-57 letters) | 15 | 8 | 23
  20/63 (58-62 letters) | 20 | 6 | 26
  20/50 (63-67 letters) | 14 | 13 | 27
Visual Acuity in the Amblyopic Eye at Randomization [Mean (Standard Deviation); unit: letters] | 52.8 (9.8) | 51.7 (11.9) | 52.4 (10.5)
Visual Acuity in the Fellow Eye at Randomization [Number; unit: participants]
  20/25 (78-82 letters) | 15 | 4 | 19
  20/20 (83-87 letters) | 35 | 20 | 55
  20/16 (88-92 letters) | 34 | 23 | 57
  20/12 (93-97 letters) | 6 | 2 | 8
Visual Acuity in the Fellow Eye at Randomization [Mean (Standard Deviation); unit: letters] | 86.7 (4.1) | 87.3 (3.5) | 86.9 (3.9)
Intraocular Visual Acuity Difference at Randomization [Mean (Standard Deviation); unit: letters] | 33.9 (10.9) | 35.6 (13.1) | 34.5 (11.7)
SE Refractive Error in Amblyopic Eye at Randomization [Mean (Standard Deviation); unit: diopters] | 4.0 (2.6) | 4.5 (2.3) | 4.2 (2.5)
SE Refractive Error in Fellow Eye at Randomization [Mean (Standard Deviation); unit: diopters] | 1.9 (2.0) | 1.6 (1.7) | 1.8 (1.9)
Anisometropia at Randomization [Mean (Standard Deviation); unit: diopters] | 2.5 (2.1) | 3.1 (2.0) | 2.7 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Distribution of Amblyopic Eye Visual Acuity Change From Baseline
Description: The primary outcome is the amblyopic eye visual acuity letter score measured at the 18-week primary outcome visit following a rapid taper of study medicine beginning at week 16. The primary analytic approach will be a treatment group comparison of the mean amblyopic eye visual acuity adjusted for baseline acuity.
  Visual acuity was measured in each eye (right eye first) by a study-certified VA tester using the Electronic Early Treatment of Diabetic Retinopathy Study (E-ETDRS©) visual acuity protocol. Five letters is equivalent to one logMAR line.
Time Frame: 18 weeks after enrollment
Population: The ITT principle was followed. For subjects with no visit in the +/- 1 wk window for the 18-wk visit, data from a visit 14-27 wks after randomization were used, if available. Multiple imputation by the Monte Carlo Markov Chain method was used for missing 18-wk VA outcomes based on tx group, baseline VA, & VA scores from completed follow-up visits.
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
participants
  10-14 letters worse | 0 | 0
  5-9 letters worse | 2 | 1
  within 4 letters | 35 | 23
  5-9 letters better | 36 | 19
  10-14 letters better | 10 | 1
  >= 15 letters better | 3 | 1

2. Secondary Outcome: Amblyopic Eye Visual Acuity Improvement Treatment Group Comparison at 18 Weeks
Description: Treatment group comparisons of the proportion of subjects who have improved from baseline by 10 or more letters.
Time Frame: 18 weeks after enrollment
Population: The analysis followed the intent-to-treat principle. For missing primary outcome visits (±1 wk), data from a visit 14-27 wks after randomization were used, if available.Multiple imputation(Monte Carlo Markov Chain method) was used for missing 18-wk VA outcomes based on treatment group, baseline VA, and VA scores from completed follow-up visits
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
participants | 13 | 2
Statistical Analysis 1: Comparison: Levodopa/Carbidopa vs Placebo; A sample size of 129 participants provided 80% power with 1-sided type I error rate of 5% to reject the hypothesis of no difference between groups if the proportion improved was 30% in the levodopa group compared with 10% in the placebo group; Test type: Superiority or Other; p = 0.06, Fisher Exact; It was not possible to adjust for baseline VA in these secondary analyses due to the small number of subjects meeting secondary outcome criteria; Percent Difference = 11, 95% CI 2-sided [-7 to 28] — Treatment group difference calculated as Levodopa - Placebo

3. Secondary Outcome: Distribution of Amblyopic Eye Visual Acuity at 18 Weeks
Time Frame: 18 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
participants
  20/25 (78-82 letters) | 0 | 0
  20/32 (73-77 letters) | 5 | 1
  20/40 (68-72 letters) | 7 | 6
  20/50 (63-67 letters) | 20 | 5
  20/63 (58-62 letters) | 18 | 9
  20/80 (53-57 letters) | 12 | 5
  20/100 (48-52 letters) | 17 | 9
  20/125 (43-47 letters) | 4 | 3
  20/160 or worse (<=42 letters) | 3 | 7

4. Secondary Outcome: Mean Amblyopic Eye Visual Acuity at 18 Weeks
Description: Visual acuity was measured in each eye (right eye first) by a study-certified VA tester using the Electronic Early Treatment of Diabetic Retinopathy Study (E-ETDRS©) visual acuity protocol. Five letters is equivalent to one logMAR line.
Time Frame: 18 weeks after enrollment
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
letters | 58.7 (8.9) | 54.8 (12.3)

5. Secondary Outcome: Amblyopic Eye Visual Acuity Improvement Treatment Group Comparison at 4 Weeks
Description: Treatment group comparisons adjusted for baseline acuity scores using logistic regression of the proportion of subjects who have improved from baseline by 10 or more letters.
Time Frame: 4 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 88 | 47
participants
  Improved 10 or more letters | 4 | 2
  Did not improve 10 or more letters | 84 | 45
Statistical Analysis 1: Comparison: Levodopa/Carbidopa vs Placebo; Test type: Superiority or Other; Percent Difference = 0, 95% CI 2-sided [-17 to 18] — Levodopa - Placebo

6. Secondary Outcome: Amblyopic Eye Visual Acuity Improvement Treatment Group Comparison at 10 Weeks
Description: Treatment group comparisons of the proportion of subjects who have improved from baseline by 10 or more letters.
Time Frame: 10 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 88 | 48
participants
  Improved 10 or more letters | 10 | 9
  Not improved 10 or more letters | 78 | 39
Statistical Analysis 1: Comparison: Levodopa/Carbidopa vs Placebo; Test type: Superiority or Other; Percent Difference = -7, 95% CI 2-sided [-25 to 10]

7. Secondary Outcome: Amblyopic Eye Visual Acuity Improvement Treatment Group Comparison at 16 Weeks
Description: Treatment group comparisons of the proportion of subjects who have improved from baseline by 10 or more letters.
Time Frame: 16 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 87 | 46
participants
  Improved 10 or more letters | 15 | 10
  Not improved 10 or more letters | 72 | 36
Statistical Analysis 1: Comparison: Levodopa/Carbidopa vs Placebo; Test type: Superiority or Other; Percent Difference = -5, 95% CI 2-sided [-22 to 13] — Levodopa - Placebo

8. Secondary Outcome: Amblyopic Eye Visual Acuity Improvement Treatment Group Comparison at 26 Weeks
Description: as for outcome 5
Time Frame: 26 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
participants
  Improved 10 or more letters | 17 | 5
  Not improved 10 or more letters | 69 | 40

9. Secondary Outcome: Amblyopia Resolutionat 4 Weeks
Description: Treatment group comparisons adjusted for baseline acuity scores using logistic regression of the proportion of subjects with 20/25 or better visual acuity.
Time Frame: 4 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 88 | 47
participants
  20/25 or better | 0 | 0
  20/32 or worse | 88 | 47

10. Secondary Outcome: Amblyopia Resolution at 10 Weeks
Description: as for outcome 9
Time Frame: 10 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 88 | 48
participants
  20/25 or better | 0 | 0
  20/32 or worse | 88 | 48

11. Secondary Outcome: Amblyopia Resolution at 16 Weeks
Description: as for outcome 9
Time Frame: 16 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 87 | 46
participants
  20/25 or better | 1 | 0
  20/32 or worse | 86 | 46

12. Secondary Outcome: Amblyopia Resolution at 18 Weeks
Description: as for outcome 9
Time Frame: 18 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
participants
  20/25 or better | 0 | 0
  20/32 or worse | 86 | 45

13. Secondary Outcome: Amblyopia Resolution at 26 Weeks
Description: as for outcome 9
Time Frame: 26 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
participants
  20/25 or better | 0 | 0
  20/32 or worse | 86 | 45

14. Secondary Outcome: Distribution of Amblyopic Eye Visual Acuity Change From Baseline at 4 Weeks
Description: as for outcome 4
Time Frame: 4 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 88 | 47
participants
  10-14 letters worse | 0 | 0
  5-9 letters worse | 6 | 2
  within 4 letters | 55 | 28
  5-9 letters better | 23 | 15
  10-14 letters better | 4 | 1
  >= 15 letters better | 0 | 1

15. Secondary Outcome: Mean Change in Amblyopic Eye Visual Acuity From Baseline at 4 Weeks
Description: A treatment group comparison of the mean amblyopic eye visual acuity at 4 weeks after enrollment, adjusted for baseline acuity.
Time Frame: 4 weeks after enrollment
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 88 | 47
letters | 2.2 (4.1) | 2.5 (4.7)
Statistical Analysis 1: Comparison: Levodopa/Carbidopa vs Placebo; Test type: Superiority or Other; p = 0.65, ANCOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.9 to 1.3] — Mean difference calculated as Levodopa - Placebo

16. Secondary Outcome: Distribution of Amblyopic Eye Visual Acuity Change From Baseline at 10 Weeks
Description: as for outcome 4
Time Frame: 10 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 88 | 48
participants
  10-14 letters worse | 1 | 0
  5-9 letters worse | 4 | 1
  within 4 letters | 43 | 30
  5-9 letters better | 30 | 8
  10-14 letters better | 7 | 9
  >= 15 letters better | 3 | 0

17. Secondary Outcome: Mean Change in Amblyopic Eye Visual Acuity From Baseline at 10 Weeks
Description: A treatment group comparison of the mean amblyopic eye visual acuity at 10 weeks after enrollment, adjusted for baseline acuity. Visual acuity was measured in each eye (right eye first) by a study-certified VA tester using the Electronic Early Treatment of Diabetic Retinopathy Study (E-ETDRS©) visual acuity protocol. Five letters is equivalent to one logMAR line.
Time Frame: 10 weeks after enrollment
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 88 | 48
letters | 3.8 (4.9) | 3.7 (4.9)
Statistical Analysis 1: Comparison: Levodopa/Carbidopa vs Placebo; Test type: Superiority or Other; p = 0.44, ANCOVA; Mean Difference (Net) = 0.1, 95% CI 2-sided [-1.6 to 1.8]

18. Secondary Outcome: Distribution of Amblyopic Eye Visual Acuity Change From Baseline at 16 Weeks
Description: as for outcome 4
Time Frame: 16 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 87 | 46
participants
  10-14 letters worse | 0 | 0
  5-9 letters worse | 1 | 0
  within 4 letters | 41 | 26
  5-9 letters better | 30 | 10
  10-14 letters better | 9 | 10
  >= 15 letters better | 6 | 0

19. Secondary Outcome: Mean Change in Amblyopic Eye Visual Acuity From Baseline at 16 Weeks
Description: A treatment group comparison of the mean amblyopic eye visual acuity at 16 weeks after enrollment, adjusted for baseline acuity. Visual acuity was measured in each eye (right eye first) by a study-certified VA tester using the Electronic Early Treatment of Diabetic Retinopathy Study (E-ETDRS©) visual acuity protocol. Five letters is equivalent to one logMAR line.
Time Frame: 16 weeks after enrollment
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 87 | 46
letters | 5.1 (6.3) | 4.2 (4.9)
Statistical Analysis 1: Comparison: Levodopa/Carbidopa vs Placebo; Test type: Superiority or Other; p = 0.20, ANCOVA; Mean Difference (Net) = 0.9, 95% CI 2-sided [-1.2 to 2.9]

20. Secondary Outcome: Distribution of Amblyopic Eye Visual Acuity Change From Baseline at 26 Weeks
Description: as for outcome 4
Time Frame: 26 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
participants
  5-9 letters worse | 3 | 1
  within 4 letters | 36 | 23
  5-9 letters better | 30 | 16
  10-14 letters better | 14 | 5
  >= 15 letters better | 3 | 0

21. Secondary Outcome: Mean Change in Amblyopic Eye Visual Acuity From Baseline at 26 Weeks
Description: A treatment group comparison of the mean amblyopic eye visual acuity at 26 weeks after enrollment, adjusted for baseline acuity. Visual acuity was measured in each eye (right eye first) by a study-certified VA tester using the Electronic Early Treatment of Diabetic Retinopathy Study (E-ETDRS©) visual acuity protocol. Five letters is equivalent to one logMAR line.
Time Frame: 26 weeks after enrollment
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
letters | 5.0 (5.7) | 4.2 (4.7)
Statistical Analysis 1: Comparison: Levodopa/Carbidopa vs Placebo; Test type: Superiority or Other; p = 0.17, ANCOVA; Mean Difference (Net) = 0.9

22. Secondary Outcome: Distribution of Fellow Eye Visual Acuity at 18 Weeks
Description: Similar to the analysis for the amblyopic eye, the fellow eye visual acuity will be evaluated to determine if study treatment had an adverse effect on the occluded eye. The analysis will be a treatment group comparison of the mean fellow eye visual acuity at 18 weeks after enrollment, adjusted for baseline acuity.
Time Frame: 18 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 87 | 45
participants
  20/12 (93-97 letters) | 12 | 4
  20/16 (88-92 letters) | 44 | 22
  20/20 (83-87 letters) | 22 | 16
  20/25 (78-82 letters) | 8 | 3
  20/32 (73-77 letters) | 1 | 0

23. Secondary Outcome: Mean Fellow Eye Visual Acuity at 18 Weeks
Description: as for outcome 4
Time Frame: 18 weeks after enrollment
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 87 | 45
letters | 88.1 (4.4) | 88.0 (3.2)

24. Secondary Outcome: Distribution of Fellow Eye Visual Acuity Change From Baseline at 18 Weeks
Description: as for outcome 4
Time Frame: 18 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 87 | 45
participants
  >=15 letters worse | 0 | 0
  10-14 letters worse | 0 | 0
  5-9 letters worse | 4 | 3
  within 4 letters | 68 | 39
  5-9 letters better | 15 | 3
  10-14 letters better | 0 | 0

25. Primary Outcome: Mean Amblyopic Eye Visual Acuity Change From Baseline
Description: as for outcome 1
Time Frame: 18 weeks after enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
letters | 5.2 (5.3) | 3.8 (5.0)
Statistical Analysis 1: Comparison: Levodopa/Carbidopa vs Placebo; With 129 participants, assuming a 1-sided type I error rate of 4.85%, there was 96% power to detect a difference in mean visual acuity between treatment groups at 18 weeks adjusted for baseline and for 1 interim analysis for futility if the true difference was 5 letters with SD of 7 letters and 82% power if the true difference was 3.75 letters; Test type: Superiority or Other; p = 0.06, ANCOVA — The alpha level was set to 0.0485 for the primary analysis to adjust for alpha spending of 0.015 for one interim analysis for efficacy conducted when outcome data were available for 50% of participants; Mean Difference (Net) = 1.4, 95% CI 2-sided [-0.4 to 3.3] — Mean difference calculated as Levodopa - Placebo

26. Secondary Outcome: Mean Fellow Eye Visual Acuity Change From Baseline at 18 Weeks
Description: as for outcome 4
Time Frame: 18 weeks after enrollment
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 87 | 45
letters | 1.5 (3.0) | 0.5 (3.1)

27. Secondary Outcome: Mean Child Symptom Survey Score at Enrollment
Description: A treatment group comparison of symptom survey scores at enrollment. The average of the overall item responses will be calculated and compared by treatment group with a t-test for difference in means. A higher number reflects a more negative response (5=always, 4=often, 3=sometimes, 2=rarely, 1=never).
Time Frame: At enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 90 | 49
units on a scale | 1.60 (0.37) | 1.73 (0.45)

28. Secondary Outcome: Mean Child Symptom Survey Score at 4 Weeks
Description: A treatment group comparison of symptom survey scores at the 4 week visit. The average of the overall item responses will be calculated and compared by treatment group with a t-test for difference in means. A higher number reflects a more negative response (5=always, 4=often, 3=sometimes, 2=rarely, 1=never).
Time Frame: 4 weeks after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 88 | 47
units on a scale | 1.42 (0.37) | 1.51 (0.42)

29. Secondary Outcome: Mean Child Symptom Survey Score at 10 Weeks
Description: A treatment group comparison of symptom survey scores at the 10 week visit. The average of the overall item responses will be calculated and compared by treatment group with a t-test for difference in means. A higher number reflects a more negative response (5=always, 4=often, 3=sometimes, 2=rarely, 1=never).
Time Frame: 10 weeks after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 88 | 47
units on a scale | 1.33 (0.31) | 1.42 (0.37)

30. Secondary Outcome: Mean Child Symptom Survey Score at 16 Weeks
Description: A treatment group comparison of symptom survey scores at the 16 week visit. The average of the overall item responses will be calculated and compared by treatment group with a t-test for difference in means. A higher number reflects a more negative response (5=always, 4=often, 3=sometimes, 2=rarely, 1=never).
Time Frame: 16 weeks after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 87 | 46
units on a scale | 1.25 (0.27) | 1.38 (0.36)

31. Secondary Outcome: Mean Child Symptom Survey Score at 18 Weeks
Description: A treatment group comparison of symptom survey scores at the primary outcome (18 week) visit. The average of the overall item responses will be calculated and compared by treatment group with a t-test for difference in means. A higher number reflects a more negative response (5=always, 4=often, 3=sometimes, 2=rarely, 1=never).
Time Frame: 18 weeks after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 87 | 45
units on a scale | 1.17 (0.22) | 1.28 (0.32)

32. Secondary Outcome: Mean Child Symptom Survey Score at 26 Weeks
Description: A treatment group comparison of symptom survey scores at the 26 week visit. The average of the overall item responses will be calculated and compared by treatment group with a t-test for difference in means. A higher number reflects a more negative response (5=always, 4=often, 3=sometimes, 2=rarely, 1=never).
Time Frame: 26 weeks after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
units on a scale | 1.23 (0.26) | 1.33 (0.32)

33. Secondary Outcome: Mean Parent Symptom Survey Score at Enrollment
Description: as for outcome 27
Time Frame: At enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 90 | 49
units on a scale | 1.42 (0.34) | 1.44 (0.29)

34. Secondary Outcome: Mean Parent Symptom Survey Score at 4 Weeks
Description: as for outcome 28
Time Frame: 4 weeks after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 88 | 47
units on a scale | 1.29 (0.27) | 1.26 (0.27)

35. Secondary Outcome: Mean Parent Symptom Survey Score at 10 Weeks
Description: as for outcome 29
Time Frame: 10 weeks after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 88 | 47
units on a scale | 1.22 (0.22) | 1.30 (0.25)

36. Secondary Outcome: Mean Parent Symptom Survey Score at 16 Weeks
Description: as for outcome 30
Time Frame: 16 weeks after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 87 | 46
units on a scale | 1.24 (0.27) | 1.25 (0.22)

37. Secondary Outcome: Mean Parent Symptom Survey Score at 18 Weeks
Description: as for outcome 31
Time Frame: 18 weeks after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 87 | 45
units on a scale | 1.17 (0.21) | 1.17 (0.20)

38. Secondary Outcome: Mean Parent Symptom Survey Score at 26 Weeks
Description: as for outcome 32
Time Frame: 26 weeks after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
units on a scale | 1.19 (0.24) | 1.22 (0.29)

39. Secondary Outcome: Mean Systemic Adverse Events
Time Frame: Enrollment through 26 weeks
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 90 | 49
events | 1.28 (1.39) | 1.55 (1.90)

40. Secondary Outcome: Distribution of Fellow Eye Visual Acuity at 26 Weeks
Description: Similar to the analysis for the amblyopic eye, the fellow eye visual acuity will be evaluated to determine if study treatment had an adverse effect on the occluded eye. The analysis will be a treatment group comparison of the mean fellow eye visual acuity at 26 weeks after enrollment, adjusted for baseline acuity.
Time Frame: 26 weeks after enrollment
Population: All participants continued in the study regardless of whether they continued with study medication after the 18-week visit; 49 participants in the levodopa group and 24 participants in the placebo group continued study medication at the 18-week visit.
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
participants
  20/12 (93-97 letters) | 15 | 7
  20/16 (88-92 letters) | 34 | 22
  20/20 (83-87 letters) | 28 | 13
  20/25 (78-82 letters) | 9 | 2
  20/32 (73-77 letters) | 0 | 1

41. Secondary Outcome: Mean Fellow Eye Visual Acuity at 26 Weeks
Description: as for outcome 4
Time Frame: 26 weeks after enrollment
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
letters | 88.0 (4.5) | 88.2 (4.1)

42. Secondary Outcome: Distribution of Fellow Eye Visual Acuity Change From Baseline at 26 Weeks
Description: as for outcome 4
Time Frame: 26 weeks after enrollment
Population: as for outcome 40
Measure: Number; unit: participants
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
participants
  >=15 letters worse | 1 | 0
  10-14 letters worse | 0 | 0
  5-9 letters worse | 2 | 4
  within 4 letters | 74 | 35
  5-9 letters better | 7 | 6
  10-14 letters better | 2 | 0

43. Secondary Outcome: Mean Fellow Eye Visual Acuity Change From Baseline at 26 Weeks
Description: as for outcome 4
Time Frame: 26 weeks after enrollment
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Levodopa/Carbidopa | Placebo
Number analyzed (Participants) | 86 | 45
letters | 1.4 (3.6) | 0.8 (3.3)

ADVERSE EVENTS:
Time Frame: From enrollment to last follow-up visit (26 weeks)
Arm/Group | Levodopa/Carbidopa | Placebo
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/49
Other Adverse Events (participants affected / at risk) | 37/90 | 17/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levodopa/Carbidopa (N=90) | Placebo (N=49)
Headache (General disorders) | 18 (23) | 4 (6)
Nausea (General disorders) | 6 (7) | 6 (6)
Cough (General disorders) | 4 (4) | 3 (4)
Gastroenteritis viral (Gastrointestinal disorders) | 4 (5) | 3 (3)
Nasopharyngitis (General disorders) | 4 (4) | 4 (4)
Pharyngitis streptococcal (General disorders) | 3 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (3)
Dry eye (Eye disorders) | 0 (0) | 4 (4)
Eye irritation (Eye disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No